CLINICAL TRIAL: NCT06217653
Title: The Effect of Baby Yoga on Sleep, Maternal Attachment and Breastfeeding Self-Efficacy: Randomized Trials
Brief Title: Baby Yoga Sleep Maternal Attachment Breastfeeding
Acronym: Baby Yoga
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Halic University (Other)
Responsible Party: Principal Investigator, Fatma Şule Bilgiç, Lecturer, Halic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Yoga Çalışma
Record Dates: First submitted 2023-03-31; First posted 2024-01-22 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Maternal Behavior; Maternal Care Patterns
Keywords: Sleep; Maternal; Baby; Yoga

STUDY DESIGN:
Intervention Model Description: The study is of the randomized controlled type.
Who Masked: Investigator
Masking Description: In the study, the researcher and statistician who collected the data were blinded due to the nature of the study. In the data, groups were coded as groups A and B, and only the non-blind researcher who collected the data knew which group was the intervention or control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- İntervention (Experimental): Intervention Group: A mother-baby yoga video prepared by the researchers was sent to the mothers in the intervention group. Before the mothers yoga practice, a 10-minute training was given about mother-baby yoga. Mothers were asked to do yoga at least 3 times a week for 4 weeks. Counseling and follow-up of the process were carried out by a researcher by calling the mothers once a week.
  Mothers were asked to choose the most suitable time of the day for the baby and herself, to have the baby fed at least 45 minutes before yoga, and to practice in a calm and dim environment, listening to music or white noise of her choice. Approximately one yoga session is 20 minutes.
  It was monitored once a week for 4 weeks, a total of 4 times. Postnatal Breastfeeding Self-Efficacy Scale-Short Form, Mother-Infant Attachment Scale, and Sleep Diary were administered to mothers at each follow-up.
  Interventions: Behavioral: mother baby yoga
- Control (No Intervention): Data Collection Form, Postnatal Breastfeeding Self-Efficacy Scale-Short Form, Mother-Infant Attachment Scale, and Sleep Diary were administered to mothers.It was monitored once a week for 4 weeks, a total of 4 times. Postnatal Breastfeeding Self-Efficacy Scale-Short Form, Mother-Infant Attachment Scale, and Sleep Diary were administered to mothers at each follow-up.

INTERVENTIONS:
Behavioral: mother baby yoga — Yoga Video Content Plan
  * Mood Regulation: Abdominal/Belly Breathing
  * Warm Touch from the Heart
  * Chair Posture
  * Bucket Wrapping
  * Bukka Bukka (Heart)
  * Vortex Generation
  * Fertile Falls
  * One Hand Two Hands
  * Tiny Stretches
  * Here and Now Awareness
  * Dolphin Pose Mothers were asked to choose the most suitable time of the day for the baby and herself, to have the baby fed at least 45 minutes before yoga, and to practice in a calm and dim environment, listening to music or white noise of her choice. Approximately one yoga session is 20 minutes.
  Arms: İntervention

SUMMARY:
The randomized controlled type study was conducted with 150 mothers and mothers who gave birth in the Haseki Training and Research Hospital Postpartum Service between February and February. The mothers included in the study were randomized 1:1 into 2 groups. The mothers of the babies in the intervention group were sent a "Baby Yoga" video shot by the researchers and asked to practice them at least 3 times a week for 4 weeks. Data are obtained with Data collection form, Mother-Infant Attachment Scale, Breastfeeding Self-Efficacy Short Form and Baby Sleep Diary.

DETAILED DESCRIPTION:
This study was conducted in a randomized controlled type to examine the effect of infant yoga practiced by mothers on infants' sleep duration, maternal attachment and breastfeeding. The enrollment, assignment, follow-up and analysis steps of the trial were demonstrated using CONSORT 2018 (Updated Guidelines for Reporting Randomized Parallel Group Studies).

While the population of the study consisted of mothers and babies who gave birth in the Haseki Training and Research Hospital Obstetrics Clinic, the minimum sample number was calculated using G Power. Accordingly, it was found that the number of samples to be taken was 68 for each group, a total of 136 mothers and their babies. Considering that there would be losses, the sample was planned to be 150 mothers and their babies, 75 for each group.

Sample Selection Criteria

* Babies born at term (37-40 weeks of gestation)
* In the first postpartum week,
* Healthy and singleton newborns were included. Sample Exclusion Criteria
* Babies staying in the postnatal intensive care unit,
* The mother has a physical disability,
* The mother has a psychiatric illness,
* Being pregnant using assisted reproductive techniques,
* Not included if the mother or baby has a disability related to breastfeeding

Data Collection Tools The data of the study were obtained by using the Data Collection Form, Postnatal Breastfeeding Self-Efficacy Scale-Short Form, Mother-Infant Attachment Scale, and Sleep Diary.

Data Collection Stages Stage 1: 150 mothers and their babies who met the sample selection criteria were included in the study in the first postpartum week. Mothers were randomized into two groups as intervention and control. Data Collection Form, Postnatal Breastfeeding Self-Efficacy Scale-Short Form, Mother-Infant Attachment Scale, and Sleep Diary were administered to all mothers.

Stage 2: Intervention Group: A mother-baby yoga video prepared by the researchers was sent to the mothers in the intervention group. Before the mothers yoga practice, a 10-minute training was given about mother-baby yoga. Mothers were asked to do yoga at least 3 times a week for 4 weeks. Counseling and follow-up of the process were carried out by a researcher by calling the mothers once a week.

Yoga Video Content Plan

* Mood Regulation: Abdominal/Belly Breathing
* Warm Touch from the Heart
* Chair Posture
* Bucket Wrapping
* Bukka Bukka (Heart)
* Vortex Generation
* Fertile Falls
* One Hand Two Hands
* Tiny Stretches
* Here and Now Awareness
* Dolphin Pose Mothers were asked to choose the most suitable time of the day for the baby and herself, to have the baby fed at least 45 minutes before yoga, and to practice in a calm and dim environment, listening to music or white noise of her choice. Approximately one yoga session is 20 minutes.

Control group: Left for routine care. Stage 3: All babies and their mothers were followed up once a week for 4 weeks, a total of 4 times. Postnatal Breastfeeding Self-Efficacy Scale-Short Form, Mother-Infant Attachment Scale, and Sleep Diary were administered to mothers at each follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Babies born at term (37-40 weeks of gestation)
* In the first postpartum week,
* Healthy and singleton newborns were included.

Exclusion Criteria:

* Babies staying in the postnatal intensive care unit,
* The mother has a physical disability,
* The mother has a psychiatric illness,
* Being pregnant using assisted reproductive techniques,
* Not included if the mother or baby has a disability related to breastfeeding

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Mother
Enrollment: 150 (Actual)
Dates: Start 2023-01-20 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Maternal Attecment | 16 weeks
  Attachment level was measured with the Mother-Infant Attachment

SECONDARY OUTCOMES:
Baby Sleep | 16 weeks
  Sleep characteristics of infants were measured by means of a sleep diary
Breastfeeding Self-Efficacy | 16 Weeks
  Breastfeeding Self-Efficacy Short Form The scale was developed by McCarter-Spaulding (2001) to measure how adequately the mother perceives her milk. The Insufficient Milk Perception scale consists of a total of 6 questions and a single subdivision. The first question on the scale is whether the mother finds her milk sufficient. The first question is answered as yes or no. The other 5 questions are scored between 0-10. The given score indicates that as it approaches zero, the mother perceives her milk as inadequate, and as she approaches 10, she perceives enough. A minimum of zero points and a maximum of 50 points can be obtained from the scale. The high score indicates that milk is sufficiently perceived. The cronbach α value of the scale was found to be 0.82 by Gökçeoğlu and Küçükoğlu (2017). In this study, the cronbach α value of the scale was found to be 0.85.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University, Fatih, Istanbul, Turkey (Türkiye)